CLINICAL TRIAL: NCT06511817
Title: Myocardial Infarction With Non-obstructive Coronary Arteries: Italian Observational
Brief Title: Myocardial Infarction With Non-obstructive Coronary Arteries: Italian Study
Acronym: MINOCA-IT
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, MONTONE ROCCO ANTONIO, MD, PhD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 6472
Record Dates: First submitted 2024-07-10; First posted 2024-07-22 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: MINOCA
MeSH Terms: conditions — MINOCA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention will be performed — No intervention will be performed

SUMMARY:
Acute coronary syndromes have been extensively studied in recent decades, focusing mainly on myocardial infarctions with obstructive coronary artery disease and early revascularisation strategies. However, the extensive use of highly sensitive troponin tests and coronary angiography has revealed a substantial group of patients with myocardial infarction without significant coronary stenosis (≥50%). This group is referred to as myocardial infarction with non-obstructive coronary arteries (MINOCA). MINOCA are defined by evidence of a myocardial infarction with normal or near-normal coronary arteries on angiography, in the absence of an alternative diagnosis specific to the clinical presentation (e.g. sepsis, myocarditis, pulmonary embolism). MINOCA may present with different aetiologies, including coronary plaque rupture/erosion, epicardial or microvascular spasm and coronary embolism. Therefore, the diagnosis of MINOCA must be considered a 'working diagnosis', which not only requires but warrants further investigation to determine the underlying cause. In fact, the investigation of MINOCA is conducted on two levels, first by excluding disorders that mimic myocardial infarction and then by identifying the cause responsible for MINOCA. In order to identify the various underlying causes of MINOCA, a cardiac MRI and/or coronary vascular imaging approach with OCT or intravascular ultrasound (IVUS) and a coronary functional assessment of microvascular function, as well as the provocation of coronary spasms by acetylcholine testing are recommended. Moreover, the clear definition of the aetiology is of great importance considering the role they play in the most appropriate therapeutic choice.

Therefore, the creation of an Italian national database could implement not only the knowledge of this clinical condition but also its management and consequent prognosis.

DETAILED DESCRIPTION:
Although the prevalence of MINOCA is about 5-25% of all myocardial infarctions and the prognosis is now recognised as inauspicious, with a one-year all-cause mortality rate of 3.5%, data on the specific demographics, clinical features, etiopathogenetic factors and prognosis of MINOCA patients are still currently unavailable in Italy. The aim of this study is to assess, in a real-world setting, prevalence, demographics, possible aetiological causes and diagnostic, therapeutic and prognostic data of MINOCA patients in Italy by creating a national database with ambispectively collected data. The collection of therapeutic and management data on MINOCA in an ambispective manner - retrospective and prospective patients - will make it possible to evaluate the hospital management of MINOCA and its association with patient prognosis over time. This database will serve to determine the incidence and characteristics of this pathology. In addition, it will make it possible to evaluate the nationwide management of patients with MINOCA, thus considering both the diagnostic aspects aimed at defining the aetiology, and cascade the treatments used and the patients' outcomes. As in all observational studies, the assessment of the risk/benefit ratio of patients with myocardial infarction, the administration of medical treatment and the management of the disease and treatment-related clinical events are the responsibility of the physician treating the patient. Since the purpose of the work only involves the collection of data, participation in this research will not entail any additional risk for the patient. The collection of actual data should provide valuable information on the demographics, aetiology and prognosis of MINOCA patients.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years;
* Diagnosis of MINOCA;
* Informed consent signed by the patient or parent/guardian/legal representative.

Exclusion criteria

* Age <18 years;
* Refusal to sign written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive consenting patients over 18 years of age diagnosed with myocardial infarction according to the Fourth Universal Definition of Myocardial Infarction and undergoing diagnostic coronary angiography and without obstructive CAD (<50%) will be included in the study from university, public and private hospitals. Patients will be included in the study by evaluating both previous patients admitted within the last 2 years (from January 2021) and consecutive patients from all centres with myocardial infarction and undergoing diagnostic coronary angiography.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is to assess the incidence of MINOCA patients in Italy, expressed as 100 person-years. | up to 2 years
  incidence of MINOCA patients in Italy, expressed as 100 person-years.

SECONDARY OUTCOMES:
To assess in real-world setting the characteristics of MINOCA patients | up to 2 years
  assess MINOCA aetiology
MACE | up to 8 years
  To assess MINOCA MACE prognostic factors at 12 months followup and up to 60 months.
MINOCA re-hospitalization | up to 8 years
  To assess MINOCA re-hospitalization prognostic factors at 12 months followup and up to 60 months.
To assess change in symptoms and quality of life through a questionnaire. | up to 8 years
  Assess quality of life through Seattle Angina Questionnaire (SAQ) questionnaires
To assess change in symptoms and quality of life through a questionnaire. | up to 8 years
  Assess quality of life through Short Form Health Survey 36 (SF-36) questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Antonio Montone, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy